CLINICAL TRIAL: NCT02953964
Title: Perceptual and Semantic Memory Encoding Strategies for People With Mild Cognitive Impairment
Brief Title: Memory Encoding Strategies for People With Mild Cognitive Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Responsible Party: Principal Investigator, Karen Liu, Associate Professor, University of Western Sydney
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Memory encoding
Record Dates: First submitted 2016-09-21; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Behavioral: perceptual-based memory encoding training (Experimental): Participants receive perceptual-based memory encoding training
  Interventions: Other: Behavioral: perceptual-based memory encoding training
- Behavioral: Semantic-based memory encoding training (Experimental): Participants receive semantic-based memory encoding training
  Interventions: Other: Behavioral: semantic-based memory encoding training
- Behavioral : control group (Active Comparator): Participants receive cognitive stimulation intervention
  Interventions: Other: Behavioral: Cognitive stimulation group (control group)

INTERVENTIONS:
Other: Behavioral: perceptual-based memory encoding training — Participants are trained in the use of perceptual-based memory encoding strategies, inclusive of visual imagery and the method of loci. Visual imagery involves the creation and encoding of mental images, while the method of loci refers to linking these images with specific places to facilitate memory (Simon et al., 2012). Participants are taught to visualise performing each step of a task in a familiar environment, such as in their home (Liu et al., 2009). After participants can correctly visualise the entire task, they then progress to actually performing the task. During the intervention sessions, 2-3 tasks are covered each session, and these tasks become progressively difficult as the weeks progress. The intervention lasts for 10 weeks with one session every week. Each session runs for 90 minutes. A follow-up home training program is run once a week for 30 minutes with the participant and their care-giver.
  Arms: Behavioral: perceptual-based memory encoding training
Other: Behavioral: semantic-based memory encoding training — Participants are asked to encode the steps of a task by forming an association of the steps and sequence. Participants are trained in the use of the chunking association method and honeycomb concept and perform different tasks each week, implementing this encoding strategy (Lim et al., 2012). The chunking association method breaks down information into smaller parts and helps with the encoding and retrieval of information. The honeycomb concept allows the steps to form a story in relation to place, time, characters, problem and solution and the story is verbalised. Participants then complete the task. During the intervention sessions, 2-3 tasks are covered each session, and these tasks become progressively difficult as the weeks progress. The intervention lasts for 10 weeks with one session every week. Each session runs for 90 minutes. A follow-up home training program is run once a week for 30 minutes with the participant and their care-giver.
  Arms: Behavioral: Semantic-based memory encoding training
Other: Behavioral: Cognitive stimulation group (control group) — Participants receiving cognitive stimulation intervention. It consists of eight sessions that train participants' visual attention and memory, auditory attention and memory and their application in daily activities. Two sessions are also given which allow for participants to apply the training practically in their daily lives. The intervention lasts for 10 weeks with one session every week. Each session runs for 90 minutes. A follow-up home training program is run once a week for 30 minutes with the participant and their care-giver.
  Other Names: Cognitive stimulation group
  Arms: Behavioral : control group

SUMMARY:
The purposes of the study are:

* To evaluate the effectiveness of a perceptual-based training program in enhancing cognitive and everyday functioning of older adults with mild cognitive impairment and mild dementia
* To evaluate the effectiveness of a semantic-based training program in enhancing cognitive and everyday functioning of older adults with mild cognitive impairment and mild dementia

DETAILED DESCRIPTION:
People with dementia experience a cognitive decline that affects their functional performance. It has been identified that encoding is less effective in people with dementia. Rehabilitating at the encoding stage is, therefore, essential. A recent systematic review found that effective interventions needed to include training in individually selected memory encoding strategies. These strategies are classified as either perceptual (visual) or semantic (association) memory encoding strategies.

Based on the above literature, the chief investigator (Associate Professor Karen Liu) ran a pilot study on an integrated home and community centre cognitive training programme for 20 elderly people with memory problem using a pre-test and post-test comparison design.

Extending on the positive results, the aim of this project was to investigate the effectiveness of perceptual and semantic encoding strategies (and compare with a control intervention). It also aims to promote the understanding of memory loss and dementia and the need for early intervention for family members of the participants.

ELIGIBILITY:
Selection Criteria:

* are aged 60 or above;
* have no previous psychiatric or memory disorder history or other neurological illness;
* have Mini-mental State Examination score (MMSE) greater than or equal to 21;
* have Clinical Dementia Rating score (CDR) of 0.5 or 1 indicating very mild and mild dementia;
* do not show sign of depression with score below 9 out of 30 in the Geriatric Depression Scale;
* are able to communicate effectively;
* have family member who can participate in the study; and
* voluntarily consent to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Disability Assessment for Dementia | Within two days before the intervention and within two days after the 10-week intervention
  Change in Disability Assessment for Dementia to assess assistance required in basic daily tasks such as dressing, bathing
Change in Instrumental Activities of Daily Living Scale | Within two days before the intervention and within two days after the 10-week intervention
  Change in Instrumental Activities of Daily Living Scale to assess assistance required in instrumental daily tasks such as laundry, meal preparation

SECONDARY OUTCOMES:
Change in Cognistat | Within two days before the intervention and within two days after the 10-week intervention
  Change in Cognistat to assess general cognitive function
Change in Digit Span Test | Within two days before the intervention and within two days after the 10-week intervention
  Change in Digit Span Test to assess attention and working memory
Change in Consortium to Establish a Registry for Alzheimer's Disease | Within two days before the intervention and within two days after the 10-week intervention
  Change in Consortium to Establish a Registry for Alzheimer's Disease to assess cognitive function in verbal fluency, memory

CONTACTS AND LOCATIONS:
Locations (2):
- Western Sydney University, Penrith, New South Wales, Australia
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mraz H, Tong CY, Liu KPY. Semantic-based memory-encoding strategy and cognitive stimulation in enhancing cognitive function and daily task performance for older adults with mild cognitive impairment: A pilot non-randomised cluster controlled trial. PLoS One. 2023 Mar 27;18(3):e0283449. doi: 10.1371/journal.pone.0283449. eCollection 2023. PMID 36972279